CLINICAL TRIAL: NCT02806882
Title: Open and Exploratory Trial to Investigate the Pharmacokinetic of Ceftaroline in Patients With CSF Device
Brief Title: Penetration of Ceftaroline Into Cerebrospinal Fluid(CSF)
Acronym: Ceftaroline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chavanet AZ 2014
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Meningitis; Ventriculitis
MeSH Terms: conditions — Meningitis | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ceftaroline fosamil (Experimental): 600mg 1 hour intravenous infusion ZINFORO
  Interventions: Drug: Ceftaroline fosamil

INTERVENTIONS:
Drug: Ceftaroline fosamil — 600mg IV infusion
  Other Names: ZINFORO

SUMMARY:
Ceftaroline is a piece of new cephalosporin very active on resistant staphylococci in methicillin (SEMR: Staphylococcus Epidermidis Resistant in Methicillin, SMAR: Staphylococcus Aureus Resistant in Methicillin)and/or in vancomycin ; Ceftaroline is also very active on pneumococci resistant in penicillin and/or 3rd generation of cephalosporins.

Ceftaroline was approved by the European Medicines Agency for the treatment of complicated skin and soft tissue infections and community-acquired pneumonia.

Scientific literature describes a good efficiency in septicemy and/or SAMR endocarditis.

Besides, a study on animal shows the efficiency of ceftaroline in meningeal infections with gram-negative Bacilli.

The rationale of this study is based on the antibacterial spectra of ceftaroline that could be used for the antibacterial treatment (curative and prophylactic) of CSF shunt associated infections.

To validate this hypothesis, it is necessary to evaluate the concentration of ceftaroline in meningeal compartment after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)

  * Provision of informed consent prior to any study specific procedures
  * Female patients of childbearing potential may be entered if pregnancy testing is negative and the patient agrees to abstain from procreational sexual intercourse or must use double-barrier contraceptive measures for the duration of the study
* Presence of an indwelling external cerebrospinal fluid (CSF) access device (ventriculostomy or lumbar drain)
* Presence of inflamed meninges as a result of documented or suspected meningitis or ventriculitis. Patients with both clinical symptoms (fever, headache, meningismus, and altered mentation) and laboratory parameters (CSF leukocytosis, defined as a CSF white blood cell count [WBC] of >10 3, elevated CSF protein, defined as CSF protein of >1g/l, reduced CSF glucose, defined as CSF glucose of <0.3g/l, or a positive CSF Gram stain or culture) indicative of CNS infection were deemed to have definitive bacterial meningitis/ventriculitis. Inflamed meninges were defined as the presence of >5 leukocytes/mm3 of CSF.

Exclusion Criteria:

* Patient has documented history of hypersensitivity or allergic reaction (urticaria, angiooedema, anaphylaxis, desquamative rash) to any β-lactam antimicrobial including cephalosporins (contraindication to cephalosporins)
* Patient is pregnant or lactating and intends to continue breastfeeding
* Severe renal insufficiency defined as creatinine clearance < 50 mL/min.
* Patients with conditions known or suspected to alter pharmacokinetics (i.e., burn or cystic fibrosis patients)
* Refusal to participate
* Person not affiliated with the social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Ceftaroline serum concentration | before infusion, at 0.5h, 1h, 3h, 6h, 12h, 24h after infusion
Ceftaroline cerebrospinal fluid concentration | before infusion, at 0.5h, 1h, 3h, 6h, 12h, 24h after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France

REFERENCES:
- [Derived] Chauzy A, Nadji A, Combes JC, Defrance N, Bouhemad B, Couet W, Chavanet P. Cerebrospinal fluid pharmacokinetics of ceftaroline in neurosurgical patients with an external ventricular drain. J Antimicrob Chemother. 2019 Mar 1;74(3):675-681. doi: 10.1093/jac/dky489. PMID 30535190